CLINICAL TRIAL: NCT05703932
Title: Examining the Effect of Home-Based Exercise on Disease Activity in Patients With Ankylosing Spondylitis Using SIRI (Systemic Inflammatory Response Index) and SII (Systemic Inflammation Index): A Randomized Controlled Trial
Brief Title: Examining the Effect of Home-Based Exercise on Disease Activity in Patients With Ankylosing Spondylitis Using SIRI and SII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Işıl Üstün, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-01-06; First posted 2023-01-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; exercise; systemic inflammatory response index; systemic inflammation index
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): AS patients diagnosed according to ASAS criteria under pharmacological treatment using NSAID ,anti-tnf and DMARD
- Home-Based Exercise Therapy Group (Active Comparator): AS patients diagnosed according to ASAS criteria under pharmacological treatment using NSAID ,anti-tnf and DMARD ;and will take exercise program including; joint range of motion and stretching exercises for cervical, thoracic and lumbar spine, stretching for erector spina, hamstring and shoulder muscles, chest expansion, abdominal and diaphragmatic breathing exercises . Exercises will be performed at submaximal level, paying attention to blood pressure, arterial (TA) and heart rate.For the patients in the exercise group, it was planned to perform the exercise program 5 days a week in 1 set with 10 repetitions, 40 minutes/day.
  Interventions: Other: home-based exercises

INTERVENTIONS:
Other: home-based exercises — Joint range of motion and stretching exercises for cervical, thoracic and lumbar spine, stretching for erector spina, hamstring and shoulder muscles, chest expansion, abdominal and diaphragmatic breathing exercises will be applied. Exercises will be performed at submaximal level, paying attention to blood pressure, arterial (TA) and heart rate.For the patients in the exercise group, it was planned to perform the exercise program 5 days a week in 1 set with 10 repetitions, 40 minutes/day.
  Arms: Home-Based Exercise Therapy Group

SUMMARY:
The systemic inflammatory response index (SIRI) is defined as "neutrophil count × monocytes/lymphocyte counts". It has been reported that SIRI can predict survival in various types of cancer, including pancreatic cancer , gallbladder cancer , oral squamous cell carcinoma , and cervical cancer. Again, SIRI can demonstrate disease activity in patients with rheumatoid arthritis (RA), It has been reported that it can predict the development of RA-related interstitial lung disease and tumor development .

Ankylosing spondylitis management strategies should be aimed at controlling disease activity, improving spinal mobility and functional status . Treatment usually includes the use of anti-inflammatory drugs to reduce pain and stiffness, and the use of disease-modifying drugs to try to stop or prevent disease progression. Patients are also advised to exercise to maintain the mobility of the spine and peripheral joints . Studies on this subject reveal that exercise is as important as drug therapy in the treatment of AS . Again, the importance of exercise in AS was emphasized in the clinical guidelines for the treatment of AS by ASAS (The Assesment in Ankylosing Spondylitis : Working Group) and EULAR (European League Against Rheumatism) . In addition to the effects of exercise on muscle strength, joint limitations, physical performance, endurance capacity and quality of life, its anti-inflammatory effects are also known.

In this study, it was aimed to evaluate the effect of exercise therapy on disease activity in AS patients with systemic inflammatory response index (SIRI) and systemic inflammation index (SII). There is not enough evidence in the literature that systemic inflammatory response index (SIRI) and systemic inflammation index (SII) can be used in the evaluation of disease activity in AS.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is an inflammatory disease of unknown etiology characterized by chronic inflammation of the sacroiliac joints, spine and paraspinal soft tissues. Extra-articular manifestations such as anterior uveitis, inflammatory bowel disease, aortic valve disease and osteoporosis may also occur. Joint fusion and dysfunction may also be seen in progressive disease states. Inflammatory low back pain and morning stiffness are common symptoms of AS. These symptoms lead to limitation of activity and exacerbation of pain in the active phase of the disease. Therefore, evaluation of disease activity in AS is very important in terms of better understanding the pathophysiology of AS, predicting prognosis, and treatment. Currently, two non-specific inflammatory biomarkers, C-reactive protein (CRP) level and erythrocyte sedimentation rate (ESH), are frequently used to monitor disease activity of rheumatic diseases; however, these biomarkers have low sensitivity and specificity . Therefore, it is necessary to identify new indicators that more accurately reflect disease activity.

Recently, complete blood cell count parameters have emerged as useful biomarkers of many inflammatory diseases due to their availability and affordability. Previous studies have shown that platelet (PLT), neutrophil, lymphocyte cell counts, red blood distribution width (RDW), neutrophil-lymphocyte ratio (NLR) and platelet-lymphocyte ratio (PLO) are important indicators of systemic inflammation. In addition, it was found that SII (Systemic Inflammation Index), calculated by the formula "platelet count × neutrophil count/lymphocyte count", increased in active-stage AS patients compared to both the healthy control group and other AS patients in remission, and showed a positive correlation with disease activity .The systemic inflammatory response index (SIRI) is defined as "neutrophil count × monocytes/lymphocyte counts". It has been reported that SIRI can predict survival in various types of cancer, including pancreatic cancer, gallbladder cancer , oral squamous cell carcinoma , and cervical cancer. Again, SIRI can demonstrate disease activity in patients with rheumatoid arthritis (RA), It has been reported that it can predict the development of RA-related interstitial lung disease and tumor development .

Ankylosing spondylitis management strategies should be aimed at controlling disease activity, improving spinal mobility and functional status . Treatment usually includes the use of anti-inflammatory drugs to reduce pain and stiffness, and the use of disease-modifying drugs to try to stop or prevent disease progression. Patients are also advised to exercise to maintain the mobility of the spine and peripheral joints . Studies on this subject reveal that exercise is as important as drug therapy in the treatment of AS . Again, the importance of exercise in AS was emphasized in the clinical guidelines for the treatment of AS by ASAS (The Assesment in Ankylosing Spondylitis : Working Group) and EULAR (European League Against Rheumatism) . In addition to the effects of exercise on muscle strength, joint limitations, physical performance, endurance capacity and quality of life, its anti-inflammatory effects are also known.

In this study, it was aimed to evaluate the effect of exercise therapy on disease activity in AS patients with systemic inflammatory response index (SIRI) and systemic inflammation index (SII). There is not enough evidence in the literature that systemic inflammatory response index (SIRI) and systemic inflammation index (SII) can be used in the evaluation of disease activity in AS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with ankylosing spondylitis according to the modified New York criteria and/or ASAS criteria

Exclusion Criteria:

* Presence of neurological disease (Epilepsy, stroke, Parkinson's, etc.)
* Severe cardiac disease (coronary artery disease, history of myocardial infarction and angina, heart failure)
* Pacemaker users
* Patients with COPD and advanced respiratory failure
* Hypertension and diabetes that cannot be controlled with medication malignancy
* Acute or chronic infections
* Organ/System dysfunction
* History of previous upper and lower extremity orthopedic surgery
* Patients with joint prosthesis
* Insufficient cooperation
* Pregnancy
* Cognitive dysfunction
* Dementia
* Presence of psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changed BASDAI score >2 in home-based exercise group measured by BASDAI-Bath Ankylosing Spondylitis Disease Activity Index at 10 week | 10 week
  The BASDAI index consists of 6 questions about disease activity. Patients are required to answer the questions considering their last week's situation and mark an appropriate point on the 10 cm horizontal line. At the beginning and end of the 10 cm horizontal line, there are the words "not at all - very severe". The average of the 2 questions about morning stiffness will be taken, added to the total of the first 4 questions, and a combined score will be obtained by dividing by 5.A higher score indicates higher disease activity.

SECONDARY OUTCOMES:
SII-systemic inflammation index | 10 week
  systemic inflammation index (SII) is defined as "platelet count × neutrophil count/lymphocyte count"
SIRI-systemic inflammatory response index | 10 week
  The systemic inflammatory response index (SIRI) is defined as "neutrophil count × monocytes/lymphocyte counts".
BASMI-Bath Ankylosing Spondylitis Metrology Index | 10 week
  BASMI consists of five clinical measurements: cervical rotation, tragus wall distance, lumbar flexion, trunk lateral flexion and intermalleolar distance.10 is highest score and indicates worst situtation.BASMI both groups before the treatment, after 6 weeks exercise program and when the treatment ends (4 weeks after) will be compared
ASDAS-CRP-Ankylosing Spondylitis Disease Activity Score-CRP | 10 week
  The ASDAS evaluation consists of four questions to be answered by the patients and the results of the acute phase reactants CRP mg/L or ESH mm/sec . Three of the questions are some questions used in BASDAI(question 2,3,6)Patients are asked to answer these questions using a VAS on a 10 cm or 100 mm long horizontal or vertical lineThe point that patients show on the VAS is calculated in cm/mm. ASDAS-CRP/ESH will be calculated together with the CRP or ESH results in the formula.
  Mild disease activity <1.3 Moderate disease activity 1.3-2.1 High disease activity 2.1-3.5 Very high disease activity is evaluated as >3.5
BASFI-Bath Ankylosing Spondylitis Functional Index | 10 week
  BASFI includes 8 items related to daily activities and 2 items related to the patient's daily life skills. Each item is evaluated on a 10 cm visual analog scale. At the beginning and end of the scale, the words "I can do it easily - I can't" are located. The patients are asked to mark on the line, considering how difficult they have been while doing the tasks during the past week. The average of 10 scales gives the total BASFI score. The total score is between 0-10. A high score indicates poor function.
ASDAS-ESR-Ankylosing Spondylitis Disease Activity Score-ESR | 10 week
  The ASDAS evaluation consists of four questions to be answered by the patients and the results of the acute phase reactants CRP mg/L or ESH mm/sec . Three of the questions are some questions used in BASDAI(question 2,3,6)Patients are asked to answer these questions using a VAS on a 10 cm or 100 mm long horizontal or vertical lineThe point that patients show on the VAS is calculated in cm/mm. ASDAS-CRP/ESH will be calculated together with the CRP or ESH results in the formula.
  Mild disease activity <1.3 Moderate disease activity 1.3-2.1 High disease activity 2.1-3.5 Very high disease activity is evaluated as >3.5
ASQoL-Ankylosing Spondylitis Quality of Life Index | 10 week
  The scale consists of 18 sentences questioning whether the patients have limitations in activities of daily living, pain, fatigue and morning stiffness, concerns about their illness, and depressed mood. The patient will be asked to answer each question as yes or no, taking into account the latest situation. Yes 1 point, no 0 points will be recorded and the total score will be calculated.
VAS-Visual Analog Scale | 10 week
  Pain is measured by visual analog scale (VAS). The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
HAD Scale-Hospital Anxiety-Depression Scale | 10 week
  Considering the last few days, each question is scored between 0-3 for the answers of the patients who are asked to give the answer that best expresses how they feel. Questions 1, 3, 5, 7, 9, 11, 13 give anxiety scores; Questions 2, 4, 6, 8, 10, 12, 14 give depression scores. The total score is obtained by summing the scores for each question. 0-7 points will be considered normal, 8-10 points will be considered borderline, while 11 points and above will be considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Isil Ustun, Study Director
Locations (1):
- Bakırkoy Dr Sadı Konuk Hospıtal, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results of the study will be written as a manuscript. In Turkey, we do not have a system sharing data to other researchers

REFERENCES:
- [Background] Lee JH, Choi M, Rim THT, Lee SC, Lee CS. Clinical Characteristics and Prognostic Factors in Ankylosing Spondylitis Associated Uveitis. Ocul Immunol Inflamm. 2019;27(1):64-69. doi: 10.1080/09273948.2017.1359630. Epub 2017 Oct 11. PMID 29020487
- [Background] Stolwijk C, Essers I, van Tubergen A, Boonen A, Bazelier MT, De Bruin ML, de Vries F. The epidemiology of extra-articular manifestations in ankylosing spondylitis: a population-based matched cohort study. Ann Rheum Dis. 2015 Jul;74(7):1373-8. doi: 10.1136/annrheumdis-2014-205253. Epub 2014 Mar 21. PMID 24658834
- [Background] Chetrit M, Khan MA, Kapadia S. State of the Art Management of Aortic Valve Disease in Ankylosing Spondylitis. Curr Rheumatol Rep. 2020 May 14;22(6):23. doi: 10.1007/s11926-020-00898-4. PMID 32410005
- [Background] Magrey MN, Lewis S, Asim Khan M. Utility of DXA scanning and risk factors for osteoporosis in ankylosing spondylitis-A prospective study. Semin Arthritis Rheum. 2016 Aug;46(1):88-94. doi: 10.1016/j.semarthrit.2016.03.003. Epub 2016 Mar 9. PMID 27162010
- [Background] Dominguez CJ, Ugalde PF, Vilchez DR, Carretero-Dios H, Estevez EC. Positive and negative affective states and disease activity in ankylosing spondylitis. Rheumatol Int. 2015 Mar;35(3):519-24. doi: 10.1007/s00296-014-3107-y. Epub 2014 Aug 15. PMID 25123554
- [Background] Poddubnyy D, Rudwaleit M, Haibel H, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. Rates and predictors of radiographic sacroiliitis progression over 2 years in patients with axial spondyloarthritis. Ann Rheum Dis. 2011 Aug;70(8):1369-74. doi: 10.1136/ard.2010.145995. Epub 2011 May 27. PMID 21622969
- [Background] Deng J, Xu S, Gao X, Xu S, Shuai Z, Pan F. Red Cell Distribution Width and Mean Platelet Volume in Patients With Ankylosing Spondylitis: A Systematic Review and Meta-analysis. J Clin Rheumatol. 2021 Oct 1;27(7):292-297. doi: 10.1097/RHU.0000000000001174. PMID 31478944
- [Background] Sezgin M, Tecer D, Kanik A, Kekik FS, Yesildal E, Akaslan E, Yildirim G, Sahin G. Serum RDW and MPV in Ankylosing Spondylitis: Can they show the disease activity? Clin Hemorheol Microcirc. 2017;65(1):1-10. doi: 10.3233/CH-162067. PMID 27258203
- [Background] Gokmen F, Akbal A, Resorlu H, Gokmen E, Guven M, Aras AB, Erbag G, Komurcu E, Akbal E, Cosar M. Neutrophil-Lymphocyte Ratio Connected to Treatment Options and Inflammation Markers of Ankylosing Spondylitis. J Clin Lab Anal. 2015 Jul;29(4):294-8. doi: 10.1002/jcla.21768. Epub 2014 May 21. PMID 24849656
- [Background] Wu J, Yan L, Chai K. Systemic immune-inflammation index is associated with disease activity in patients with ankylosing spondylitis. J Clin Lab Anal. 2021 Sep;35(9):e23964. doi: 10.1002/jcla.23964. Epub 2021 Aug 21. PMID 34418163
- [Background] Topkan E, Mertsoylu H, Kucuk A, Besen AA, Sezer A, Sezen D, Bolukbasi Y, Selek U, Pehlivan B. Low Systemic Inflammation Response Index Predicts Good Prognosis in Locally Advanced Pancreatic Carcinoma Patients Treated with Concurrent Chemoradiotherapy. Gastroenterol Res Pract. 2020 Jul 30;2020:5701949. doi: 10.1155/2020/5701949. eCollection 2020. PMID 32802045
- [Background] Sun L, Hu W, Liu M, Chen Y, Jin B, Xu H, Du S, Xu Y, Zhao H, Lu X, Sang X, Zhong S, Yang H, Mao Y. High Systemic Inflammation Response Index (SIRI) Indicates Poor Outcome in Gallbladder Cancer Patients with Surgical Resection: A Single Institution Experience in China. Cancer Res Treat. 2020 Oct;52(4):1199-1210. doi: 10.4143/crt.2020.303. Epub 2020 Jul 21. PMID 32718144
- [Background] Lin J, Chen L, Chen Q, Zhuang Z, Bao X, Qian J, Hong Y, Yan L, Lin L, Shi B, Qiu Y, Pan L, Wei L, Zheng X, Wang J, Liu F, He B, Chen F. Prognostic value of preoperative systemic inflammation response index in patients with oral squamous cell carcinoma: Propensity score-based analysis. Head Neck. 2020 Nov;42(11):3263-3274. doi: 10.1002/hed.26375. Epub 2020 Jul 18. PMID 32681711
- [Background] Xu Y, He H, Zang Y, Yu Z, Hu H, Cui J, Wang W, Gao Y, Wei H, Wang Z. Systemic inflammation response index (SIRI) as a novel biomarker in patients with rheumatoid arthritis: a multi-center retrospective study. Clin Rheumatol. 2022 Jul;41(7):1989-2000. doi: 10.1007/s10067-022-06122-1. Epub 2022 Mar 9. PMID 35266094
- [Background] Ozdemir O. Quality of life in patients with ankylosing spondylitis: relationships with spinal mobility, disease activity and functional status. Rheumatol Int. 2011 May;31(5):605-10. doi: 10.1007/s00296-009-1328-2. Epub 2010 Jan 5. PMID 20049451
- [Background] Hidding A, van der Linden S, Boers M, Gielen X, de Witte L, Kester A, Dijkmans B, Moolenburgh D. Is group physical therapy superior to individualized therapy in ankylosing spondylitis? A randomized controlled trial. Arthritis Care Res. 1993 Sep;6(3):117-25. doi: 10.1002/art.1790060303. PMID 8130287
- [Background] Dougados M, van der Heijde D. Ankylosing spondylitis: how should the disease be assessed? Best Pract Res Clin Rheumatol. 2002 Sep;16(4):605-18. doi: 10.1053/berh.2002.0252. PMID 12406429
- [Background] Heikkila S, Viitanen JV, Kautiainen H, Kauppi M. Sensitivity to change of mobility tests; effect of short term intensive physiotherapy and exercise on spinal, hip, and shoulder measurements in spondyloarthropathy. J Rheumatol. 2000 May;27(5):1251-6. PMID 10813296
- [Background] Nolte K, van Rensburg DCJ, Fletcher L. Effects of a 6-month exercise programme on disease activity, physical and functional parameters in patients with ankylosing spondylitis: Randomised controlled trial. S Afr J Physiother. 2021 Jun 29;77(1):1546. doi: 10.4102/sajp.v77i1.1546. eCollection 2021. PMID 34230900
- [Background] Zochling J, van der Heijde D, Burgos-Vargas R, Collantes E, Davis JC Jr, Dijkmans B, Dougados M, Geher P, Inman RD, Khan MA, Kvien TK, Leirisalo-Repo M, Olivieri I, Pavelka K, Sieper J, Stucki G, Sturrock RD, van der Linden S, Wendling D, Bohm H, van Royen BJ, Braun J; 'ASsessment in AS' international working group; European League Against Rheumatism. ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2006 Apr;65(4):442-52. doi: 10.1136/ard.2005.041137. Epub 2005 Aug 26. PMID 16126791
- [Background] Machado PM, Landewe R, Heijde DV; Assessment of SpondyloArthritis international Society (ASAS). Ankylosing Spondylitis Disease Activity Score (ASDAS): 2018 update of the nomenclature for disease activity states. Ann Rheum Dis. 2018 Oct;77(10):1539-1540. doi: 10.1136/annrheumdis-2018-213184. Epub 2018 Feb 16. No abstract available. PMID 29453216